CLINICAL TRIAL: NCT00251498
Title: Phase II Study of Cetuximab in Combination With Carboplatin and Docetaxel for Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Veeda Oncology (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-04-002
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Metastatic 1st line NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Cycle 1:400 mg/m2, administered as a 120-minute iv infusion on Day 1 and 250 mg/m2 administered as a 60-minute iv infusion on Days 8 and 15, subsequent cycles:250 mg/m2 administered as a 60-minute iv infusion on Days 1, 8, 15

SUMMARY:
The primary objective of this study is to determine the efficacy (response rate) of cetuximab when administered in combination with docetaxel and carboplatin for treatment of patients with advanced non-small cell lung cancer.

The secondary objectives of this study are:

* to determine the time to progression and overall survival for patients with advanced NSCLC who are treated with the combination docetaxel, carboplatin , and cetuximab
* to determine the toxicity of the combination in patients with advanced NSCLC.

Patients with stages IIIB (pleural or pericardial effusion) and IV NSCLC who have not received any prior chemotherapy will be eligible to participate in the trial. Other eligibility criteria include: ECOG PS 0-1, normal hepatic and renal function, age >18 years. Specific inclusion and exclusion criteria are detailed in Sections 4.2 and 4.3.

DETAILED DESCRIPTION:
This is a phase II, open label, non-randomized study in patients with histologically/cytologically confirmed stage IIIB (pleural or pericardial effusion) or stage IV NSCLC who have not received prior chemotherapy. The trial will evaluate the efficacy and safety profile of the combination of docetaxel, carboplatin and cetuximab for patients with advanced NSCLC.

Patients will receive a combination of docetaxel and carboplatin administered every 3 weeks plus cetuximab given weekly. A maximum of four cycles of chemotherapy will be administered to patients. Patients who demonstrate an ongoing response (CR/PR/SD) at the end of 4th cycle of chemotherapy, may receive two more cycles of treatment. Patients who continue to respond (CR/PR/SD) after six cycles of therapy may receive therapy with single agent cetuximab (250 mg/m2/week) for up to 1 year or until disease progression or unacceptable toxicity, whichever occurs first.

Patients will be evaluated for response, time to progression, and overall survival. In addition, the safety profile of the combination will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed stage IIIB (pleural or pericardial effusion) or stage IV NSCLC.
* Age > 18 years.
* ECOG PS 0-1.
* No prior chemotherapy for NSCLC.
* Measurable disease by RECIST criteria.
* Signed IRB-approved informed consent.
* Adequate bone marrow function defined by: peripheral absolute neutrophil count (ANC) >1500/microL, hemoglobin >9.0 g/dL, and platelet count >100,000/microL.
* Adequate renal function as defined by serum creatinine level less than institutional upper limit of normal (ULN) or calculated/measured creatinine clearance > 65 mL/min.
* Adequate liver function defined as: serum total bilirubin <ULN, serum aspartate aminotransferase (AST) <2.5 times ULN.
* Estimated life expectancy >12 weeks.

Exclusion Criteria:

* Untreated clinically active brain metastasis.
* Radiotherapy within 2 weeks prior to registration or previous irradiation to the only area of measurable disease.
* Treatment with any investigational therapy within 4 weeks prior to registration.
* Prior therapy with an agent that is known to specifically and directly target the EGFR pathway.
* History of any cancer other than NSCLC (except non-melanoma skin cancer or carcinoma in situ of the cervix) within the last 5 years.
* Patients in their reproductive age group should consent to use an effective method of birth control while on treatment and for at least 3 months thereafter. Patients who are breast-feeding, or have a positive pregnancy test will be excluded from the study.
* Major surgery within 3 weeks prior to registration.
* Use of immunosuppressive agents including systemic corticosteroids within 4 weeks prior to registration (corticosteroids are permitted as physiological replacement therapy or as supportive care for nausea and emesis).
* Known history of human immunodeficiency virus infection.
* Any co-morbidity or condition of sufficient severity to limit full compliance with the protocol per assessment by the investigator.
* Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction.
* Concurrent serious infection.
* History of known hypersensitivity to docetaxel or other drugs formulated with polysorbate 80.
* History of prior severe infusion reaction to a monoclonal antibody.
* Patient has >Grade 2 peripheral neuropathy within 14 days prior to registration

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Belani, MD, Principal Investigator — Veeda Oncology
Locations (1):
- Veeda Oncology, Houston, Texas, United States